CLINICAL TRIAL: NCT00993096
Title: A Trial Investigating the Pharmacodynamic Response of NN5401 in Subjects With Type 1 Diabetes
Brief Title: Investigation of the Response Relationship of NN5401 in Type 1 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-3539; 2008-008472-14 (EudraCT Number); U1111-1111-9032 (Other: WHO)
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec, insulin aspart drug combination; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- IDegAsp low (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- IDegAsp middle (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- IDegAsp high (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- BIAsp 30 low (Experimental)
  Interventions: Drug: biphasic insulin aspart 30
- BIAsp 30 middle (Experimental)
  Interventions: Drug: biphasic insulin aspart 30
- BIAsp 30 high (Experimental)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Single dose of 0.4 U/kg body weight injected subcutaneously (under the skin)
  Arms: IDegAsp low
Drug: insulin degludec/insulin aspart — Single dose of 0.6 U/kg body weight injected subcutaneously (under the skin)
  Arms: IDegAsp middle
Drug: insulin degludec/insulin aspart — Single dose of 0.8 U/kg body weight injected subcutaneously (under the skin)
  Arms: IDegAsp high
Drug: biphasic insulin aspart 30 — Single dose of 0.4 U/kg body weight injected subcutaneously (under the skin)
  Arms: BIAsp 30 low
Drug: biphasic insulin aspart 30 — Single dose of 0.6 U/kg body weight injected subcutaneously (under the skin)
  Arms: BIAsp 30 middle
Drug: biphasic insulin aspart 30 — Single dose of 0.8 U/kg body weight injected subcutaneously (under the skin)
  Arms: BIAsp 30 high

SUMMARY:
This trial was conducted in Europe. The aim of this clinical trial was to evaluate the pharmacodynamic dose-response relationship of NN5401 (insulin degludec/insulin aspart) at three therapeutically relevant doses in subjects with type 1 diabetes.

The trial is designed as a four period, incomplete block cross-over trial where the trial participant will be randomised to a treatment sequence by which the subject will receive two matched dose levels of NN5401 and biphasic insulin aspart, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Supine blood pressure at screening (after resting for 5 min) outside the range of 90-140 mmHg for systolic or 50-90 mmHg for diastolic
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Area (AUC) under the glucose infusion rate curve | From 0 to 24 hours after single-dose administration

SECONDARY OUTCOMES:
Area (AUC) under the insulin aspart concentration time curve | From 0 to 24 hours after single-dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Nosek L, Klein O, Coester H, Svendsen AL, Haahr H. Insulin degludec/insulin aspart produces a dose-proportional glucose-lowering effect in subjects with type 1 diabetes mellitus. Diabetes Obes Metab. 2015 Jul;17(7):659-64. doi: 10.1111/dom.12463. Epub 2015 May 1. PMID 25772444
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com